CLINICAL TRIAL: NCT06802224
Title: Norepinephrine vs Phenylephrine as the First-line Vasopressor to Prevent Postoperative Acute Kidney Injury After Major Non-cardiac Surgery
Brief Title: The Choice of Vasopressor to Prevent Postoperative Acute Kidney Injury After Major Non-Cardiac Surgery
Acronym: VEGA-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other); Henry Ford Health System (Other); University of Washington (Other); University of Texas Southwestern Medical Center (Other); Wake Forest University Health Sciences (Other); University of Virginia (Other); University of Maryland (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-39683; R01DK139484 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-01-31 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Surgery With General Anesthesia; Noncardiac Surgery; Hypotension During Surgery; Acute Kidney Injury (AKI); Myocardial Injury After Noncardiac Surgery (MINS); Vasopressor
Keywords: Norepinephrine; Phenylephrine; Major adverse kidney events; Pragmatic; Cluster randomized; Crossover
MeSH Terms: conditions — Acute Kidney Injury | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, multiple periods, cluster-randomized, crossover trial design in 10 to 12 sites of the Multicenter Perioperative Outcomes Group (MPOG). The randomization at each site will alternate on a monthly basis between the norepinephrine arm and phenylephrine arm. Each cluster will be a different medical center in a different health system in North America. There will be a 2 month run-in at each site, followed by 12 crossover periods with data collection (6 months randomized to PE, 6 months randomized to NE).
  This cluster randomization aligns with current clinical practice and is therefore more feasible than an individualized randomization. It also enrolls a diverse population representative of the population being treated in the participating centers. This cluster-randomized crossover design increases the power and the ability to show a realistic difference between the two groups through enrollment of a very large number of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norepinephrine (Active Comparator): Norepinephrine as the first-line intraoperative vasopressor during general anesthesia.
  Interventions: Drug: Norepinephrine
- Phenylephrine (Active Comparator): Phenylephrine as the first-line intraoperative vasopressor during general anesthesia
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — Intravenous Norepinephrine for both infusion and bolus dosing
  Arms: Norepinephrine
Drug: Phenylephrine — Intravenous Phenylephrine for both infusion and bolus dosing
  Arms: Phenylephrine

SUMMARY:
Low blood pressure, also known as hypotension, is very common during major surgery under general anesthesia. Prolonged or severe hypotension can lead to complications such as kidney injury after surgery that slow down patient recovery. Anesthesiologists commonly administer medications called vasopressors to treat low blood pressure during surgery. These medications help raise the blood pressure back up to a safe range. Two vasopressor medications are commonly used for this purpose: norepinephrine and phenylephrine. Each of these medications has slightly different effects on the heart and blood vessels (cardiovascular system). It remains unknown which of these standard medications is better for treating low blood pressure during surgery. The goal of this clinical trial is to determine which of these two medications is better at preventing injury to the kidneys after major noncardiac surgery as well as other complications such as heart problems. Major surgeries are defined as those lasting at least two hours under general anesthesia. This trial will randomize about ten centers in North America to use either norepinephrine or phenylephrine as the primary medication to treat low blood pressure in adults undergoing major noncardiac surgery. Each hospital will prioritize one of the drugs each month, and the assigned drug will rotate each month at each hospital. No further participant involvement will be required as de-identified data are collected as part of standard medical care.

DETAILED DESCRIPTION:
VEGA-2 is an open-label, pragmatic, multiple periods, cluster-randomized, crossover trial across hospitals from MPOG. Hospital centers will be assigned to use either phenylephrine (PE) or norepinephrine (NE) for the first-line intravenous vasopressor in the operating room for the treatment of intraoperative hypotension. Centers will be randomly assigned to use PE during even-numbered months and NE during odd-numbered months, or vice versa. Data will be collected from routine clinical care and automatically extracted from the electronic health record. No additional lab tests or procedures will be required for the study. Only the randomization (of each hospital to the sequence of interventions) will be different from usual care.

The intervention is the first line vasopressor used for both infusion and bolus dosing, either PE or NE . Anesthesia providers will use the concentration that their respective center already uses in line with local anesthesia and pharmacy standard operating procedures. Anesthesiologists will provide standard of care during the intraoperative period. They will evaluate the need for vasopressors based on hemodynamic assessment and the arterial pressure goals during the procedure. Anesthesia providers will be encouraged to maintain mean arterial pressure above 65 mmHg or within 20% from baseline, but the arterial pressure targets can be adjusted on an individual basis, for instance during pre-surgical time-out, or based on individual assessment. Doses of bolus or continuous infusion of vasopressors will be adjusted to reach these goals on an individual basis. Of note, the anesthesia provider could use the alternative vasopressor if they consider the benefit of one drug being higher. A second line vasopressor will be allowed. The choice of the first line vasopressors will be determined by the randomization block.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Surgery under general anesthesia with a surgery duration of 2 hours or more
* Received intravenous vasopressors during surgery

Exclusion Criteria:

* Cardiac surgery
* Extra-corporeal membrane oxygenation
* Organ transplantation
* Obstetric procedures
* Procedures on the kidney
* Outpatient procedures
* Already receiving NE or PE or inotropes before induction of anesthesia (at the time of anesthesia start)
* American Society of Anesthesiologists physical status classification 5 or 6
* Patient for whom a local protocol recommends a specific first line vasopressor
* Most recent documented estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73m^2 or preoperative renal replacement therapy within 60 days before surgery
* Patients who do not have a preoperative creatinine value within 60 days before surgery
* Alive patients who do not have a postoperative creatinine value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) | 7 days
  AKI will be defined by the change of serum creatinine based on the Kidney Disease Improving Global Outcomes (KDIGO) criteria.

SECONDARY OUTCOMES:
Major Adverse Kidney Events (MAKE) | 28 days
  The composite of severe AKI (i.e. stage 2 or 3 AKI based on the KDIGO creatinine-based definition), absence of renal recovery, and/or death.

OTHER OUTCOMES:
Myocardial Injury after Noncardiac Surgery (MINS) | 28 days
  Elevated cardiac normal or high-sensitivity troponin.
Hospital length of stay | 28 days
  Number of days of inpatient admission.
Hypotension | During anesthesia care
  Mean arterial pressure less than 65 mmHg for at least 15 cumulative minutes.
Duration of hypotension | During anesthesia care
  The cumulative number of minutes with mean arterial pressure less than 65 mmHg.
Severe hypotension | During anesthesia care
  Mean arterial pressure less than 55 mmHg for at least 15 cumulative minutes.
Duration of severe hypotension | During anesthesia care
  The cumulative number of minutes with mean arterial pressure less than 55 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Kheterpal, MD MBA, Principal Investigator — University of Michigan; Matthieu Legrand, MD PhD, Principal Investigator — University of California, San Francisco; Allison Janda, MD, Study Director — University of Michigan; Michael P Bokoch, MD PhD, Study Director — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu C, Fong N, Lazzareschi D, Mavrothalassitis O, Kothari R, Chen LL, Pirracchio R, Kheterpal S, Domino KB, Mathis M, Legrand M. Fluids, vasopressors, and acute kidney injury after major abdominal surgery between 2015 and 2019: a multicentre retrospective analysis. Br J Anaesth. 2022 Sep;129(3):317-326. doi: 10.1016/j.bja.2022.05.002. Epub 2022 Jun 8. PMID 35688657
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Pancaro C, Shah N, Pasma W, Saager L, Cassidy R, van Klei W, Kooij F, Vittali D, Hollmann MW, Kheterpal S, Lirk P. Risk of Major Complications After Perioperative Norepinephrine Infusion Through Peripheral Intravenous Lines in a Multicenter Study. Anesth Analg. 2020 Oct;131(4):1060-1065. doi: 10.1213/ANE.0000000000004445. PMID 32925324
- [Background] Prowle JR, Forni LG, Bell M, Chew MS, Edwards M, Grams ME, Grocott MPW, Liu KD, McIlroy D, Murray PT, Ostermann M, Zarbock A, Bagshaw SM, Bartz R, Bell S, Bihorac A, Gan TJ, Hobson CE, Joannidis M, Koyner JL, Levett DZH, Mehta RL, Miller TE, Mythen MG, Nadim MK, Pearse RM, Rimmele T, Ronco C, Shaw AD, Kellum JA. Postoperative acute kidney injury in adult non-cardiac surgery: joint consensus report of the Acute Disease Quality Initiative and PeriOperative Quality Initiative. Nat Rev Nephrol. 2021 Sep;17(9):605-618. doi: 10.1038/s41581-021-00418-2. Epub 2021 May 11. PMID 33976395
- [Background] Mets B. Should Norepinephrine, Rather than Phenylephrine, Be Considered the Primary Vasopressor in Anesthetic Practice? Anesth Analg. 2016 May;122(5):1707-14. doi: 10.1213/ANE.0000000000001239. No abstract available. PMID 27101504
- [Background] Legrand M, Zarbock A. Ten tips to optimize vasopressors use in the critically ill patient with hypotension. Intensive Care Med. 2022 Jun;48(6):736-739. doi: 10.1007/s00134-022-06708-y. Epub 2022 May 3. No abstract available. PMID 35504977
- [Background] Mathis MR, Naik BI, Freundlich RE, Shanks AM, Heung M, Kim M, Burns ML, Colquhoun DA, Rangrass G, Janda A, Engoren MC, Saager L, Tremper KK, Kheterpal S, Aziz MF, Coffman T, Durieux ME, Levy WJ, Schonberger RB, Soto R, Wilczak J, Berman MF, Berris J, Biggs DA, Coles P, Craft RM, Cummings KC, Ellis TA 2nd, Fleishut PM, Helsten DL, Jameson LC, van Klei WA, Kooij F, LaGorio J, Lins S, Miller SA, Molina S, Nair B, Paganelli WC, Peterson W, Tom S, Wanderer JP, Wedeven C; Multicenter Perioperative Outcomes Group Investigators. Preoperative Risk and the Association between Hypotension and Postoperative Acute Kidney Injury. Anesthesiology. 2020 Mar;132(3):461-475. doi: 10.1097/ALN.0000000000003063. PMID 31794513
- [Background] Salmasi V, Maheshwari K, Yang D, Mascha EJ, Singh A, Sessler DI, Kurz A. Relationship between Intraoperative Hypotension, Defined by Either Reduction from Baseline or Absolute Thresholds, and Acute Kidney and Myocardial Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2017 Jan;126(1):47-65. doi: 10.1097/ALN.0000000000001432. PMID 27792044
- [Background] Legrand M, Kothari R, Fong N, Palaniappa N, Boldt D, Chen LL, Kurien P, Gabel E, Sturgess-DaPrato J, Harhay MO, Pirracchio R, Bokoch MP; VEGA-1 trial investigators. Norepinephrine versus phenylephrine for treating hypotension during general anaesthesia in adult patients undergoing major noncardiac surgery: a multicentre, open-label, cluster-randomised, crossover, feasibility, and pilot trial. Br J Anaesth. 2023 May;130(5):519-527. doi: 10.1016/j.bja.2023.02.004. Epub 2023 Mar 14. PMID 36925330